CLINICAL TRIAL: NCT00759226
Title: An Open Labeled Phase 2 Study of Gemcitabine in Combination With Cisplatin, 5-FU (24h CI) and Folinic Acid in Patients With Inoperable Esophageal Cancer
Brief Title: Chemotherapeutic Trial With Gemcitabine, Cisplatin, 5-FU and Folinic Acid in Esophageal Cancer
Acronym: CONKO-101
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CONKO-Studiengruppe (Other)
Collaborators: Eli Lilly and Company (Industry); medac GmbH (Industry)
Responsible Party: Prof. Hanno Riess, Dr. Helmut Oettle, Charite Universitätsmedizin Berlin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CONKO-101
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2008-09

CONDITIONS: Esophageal Cancer
Keywords: esophageal cancer; Gemcitabine; Cisplatin; 5-FU; Folinic Acid; inoperable esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Gemcitabine; Cisplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine 1000 mg/m2 (30 min)
  Other Names: Gemzar
Drug: Cisplatin — Cisplatin 30 mg/m2 (90 min)
  Other Names: Cisplatin medac
Drug: 5-FU — 5-FU 750 mg/m2 (24h CI)
  Other Names: 5-FU medac
Drug: Folinic Acid — Folinic Acid 200 mg/m2 (30 min)
  Other Names: Rescuvolin

SUMMARY:
This multicenter open labeled phase 2 trial examines the efficacy of a combination of Gemcitabine 1000 mg/m2 (30 min), Cisplatin 30 mg/m2 (90 min), Folinic Acid 200 mg/m2 (30 min) and 5-FU 750 mg/m2 (24h CI) all given day 1,8 q D22 in patients with inoperable esophageal cancer. The combination was considered to be suitable for further evaluation with a freedom of progression rate (PR+CR+SD) of more than 60% and not be be of further interest with a rate of less than 40%. Given an alpha error of 5% and an beta error of 10% at least 66 evaluable patients were needed based on a 2-Stage Simon design with a first evaluation after 25 evaluable patients.

ELIGIBILITY:
Inclusion Criteria:

* Age>=18
* Histologically proven inoperable esophageal cancer
* Karnofsky Performance status >=60%
* Estimated life expectancy of > 12 weeks
* Measurable disease
* No other oncologic therapy
* Measurable disease
* Adequate bone marrow function
* Geographic proximity and compliance
* Informed consent
* Negative pregnancy test and adequate contraception

Exclusion Criteria:

* Insufficient hepatic or renal function
* Elevated serum calcium
* Pregnancy/breast feeding
* Active infection
* Other malignancies
* Systemic tumour complications requiring emergency interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2002-07; Primary Completion 2005-07 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Primary endpoint rate of freedom of progression (PR+CR+SD). | Max. 8 cycles of therapy

SECONDARY OUTCOMES:
Secondary endpoint median survival, progression free survival and toxicity. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Hanno Riess, MD, PhD, Principal Investigator — Charite Universitätsmedizin Berlin
Locations (1):
- Charite Universitätsmedizin Berlin, Berlin, Germany